CLINICAL TRIAL: NCT05491369
Title: Effectiveness of an Epilepsy Educational Application for Self-management in Viet Nam: a Randomized Clinical Trial
Brief Title: Effectiveness of an Epilepsy Application for Self-management in Viet Nam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Minh-An Thuy Le, Lecturer, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22416 - ĐHYD
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; Self-management; Mobile health application; Effectiveness
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial (RCT): parallel, two-arm design
Who Masked: Participant, Outcomes Assessor
Masking Description: In an attempt to blind the participants, they will be told there will be two start times for using the app, with randomization to either date. The outcome assessor will not know which group participants are in
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application users (Active Comparator): Participants will use application for self-management.
  Interventions: Other: Epilepsy application
- Control group (No Intervention): Participants will be in the waiting list which don't use the app.

INTERVENTIONS:
Other: Epilepsy application — Nanacara is an epilepsy application which helps people with epilepsy to self-manage their conditions.
  Arms: Application users

SUMMARY:
Epilepsy is a common neurological disease which effects all genders, ages and geographic regions. Self-management refers to "the ability of the individual, in conjunction with family, community, and healthcare professionals, to manage symptoms, treatments, lifestyle changes, and psychosocial, cultural, and spiritual consequences of health conditions". Optimal self-management may improve self-efficacy, knowledge about epilepsy of people with epilepsy (PWE) and family, medical compliance and avoidance of seizure triggers. This study aims to determine the effectiveness of the epilepsy app for PWE to improve self-management

DETAILED DESCRIPTION:
Epilepsy which affects over 70 million people worldwide, is one of the most common neurological diseases. Epilepsy is "a disease characterized by an enduring predisposition to generate epileptic seizures and by the neurobiological, cognitive, psychological, and social consequences of this condition." Therefore, self-management plays a crucial role for people with epilepsy (PWE) to adapt their lifestyles and behaviors for those long-lasting changes. Self-management is a dynamic, interactive, and daily process in which individuals engage to manage a chronic illness. Self-management is "the ability of the individual, in conjunction with family, community, and healthcare professionals, to manage symptoms, treatments, lifestyle changes, and psychosocial, cultural, and spiritual consequences of health conditions." Optimal self-management may improve self-efficacy, knowledge about epilepsy of PWE and family, medical compliance, and avoidance of seizure triggers.

Mobile health (mHealth) epilepsy application (apps) refers to any digital software (e.g., via the Internet, mobile device, wearable, or desktop platforms) capable of collecting, tracking, or sharing data while interacting with patients about their epilepsy health information. Recent studies have reported that mHealth applications improved the management of people with chronic illnesses, including epilepsy. In the digital era, smartphones are becoming more and more popular worldwide. In 2016, there were 24.8 million (30% of the population) smartphone users in Viet Nam, and this share is predicted to rise by 40 percent by 2021. Nanacara is an educational app for PWE to improve self-management.

A systematic review showed 20 English apps designed to improve self-management for PWE. Only one randomized clinical trial (RCT) study showed the effectiveness of mobile apps in increasing self-management for PWE. This result implied the lack of validation study related to the clinical use of the epilepsy apps. This study aims to determine the effectiveness of the epilepsy app for PWE to improve self-management.

ELIGIBILITY:
Inclusion Criteria:

* People with epilepsy diagnosed and treated by neurologists
* Smartphone users

Exclusion Criteria:

* Substance dependence
* Suicidality
* Limited language proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Epilepsy Self-Management Scale (ESMS) | 3-month
  The ESMS (DiIorio et al., 2004) is a 38-item scale categorized into 5 domains: information, medication, seizure, safety and lifestyle management. Higher scores indicate more frequent use of self-management strategies.
Quality of Life in Epilepsy Inventory (QOLIE-31) | 3-month
  The QOLIE-31 reflects the patient's subjective well-being toward his or her QOL in various aspects related to epilepsy, with higher scores indicating better wellbeing.

SECONDARY OUTCOMES:
PHQ9 (Patient Health Questionnaire scale) | 3-month
  PHQ9 is a self-reported questionnaire to assess depression.
GAD7 (Generalized Anxiety Disorder scale) | 3-month
  Assess generalized anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Minh-An T Le, Master, Study Chair — University of Medicine and Pharmacy at HCMC
Locations (2):
- Vietnam (2):
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City
  - University Medical Center at Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yoo S, Lim K, Baek H, Jang SK, Hwang GY, Kim H, Hwang H. Developing a mobile epilepsy management application integrated with an electronic health record for effective seizure management. Int J Med Inform. 2020 Feb;134:104051. doi: 10.1016/j.ijmedinf.2019.104051. Epub 2019 Dec 4. PMID 31837500
- [Result] Pandey DK, Dasgupta R, Levy J, Wang H, Serafini A, Habibi M, Song W, Shafer PO, Loeb JA. Enhancing epilepsy self-management and quality of life for adults with epilepsy with varying social and educational backgrounds using PAUSE to Learn Your Epilepsy. Epilepsy Behav. 2020 Oct;111:107228. doi: 10.1016/j.yebeh.2020.107228. Epub 2020 Jun 27. PMID 32599431
- [Result] Le Marne FA, Butler S, Beavis E, Gill D, Bye AME. EpApp: Development and evaluation of a smartphone/tablet app for adolescents with epilepsy. J Clin Neurosci. 2018 Apr;50:214-220. doi: 10.1016/j.jocn.2018.01.065. PMID 29422360
- [Result] Si Y, Xiao X, Xia C, Guo J, Hao Q, Mo Q, Niu Y, Sun H. Optimising epilepsy management with a smartphone application: a randomised controlled trial. Med J Aust. 2020 Apr;212(6):258-262. doi: 10.5694/mja2.50520. Epub 2020 Feb 24. PMID 32092160